CLINICAL TRIAL: NCT02340325
Title: The Safety of Topically Delivered FS2 in Humans. Phase 1 Clinical Trial
Brief Title: FS2 Safety and Tolerability Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: British Columbia Professional Firefighters' Burn and Wound Healing Laboratory (Other)
Responsible Party: Principal Investigator, Anthony Papp, Medical Director, British Columbia Professional Firefighters' Burn and Wound Healing Laboratory
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: H14-00143
Record Dates: First submitted 2014-12-01; First posted 2015-01-16 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Cicatrix; Cicatrix, Hypertrophic; Keloid
MeSH Terms: conditions — Cicatrix; Cicatrix, Hypertrophic; Keloid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acute Sensitivity Test to FS2 cream (Other): Twenty (20) healthy volunteers will be assigned volunteer numbers and will have a testing areas identified by permanent marker on their backs. Pouches containing 0.00% (placebo), 0.15%, 0.25%, 0.4% and 0.5% of FS2 will be randomly applied to an occlusive, transparent dressing (Tegaderm) and applied to each test area once for 24 hours. The pouch order will be random, generated by the www.random.org list generator each application. Patients will be evaluated at 24 hours post application for skin reactions and adverse reactions by a blinded observer recorded. Before and after photographs will be taken.
  Interventions: Drug: Acute Application of kynurenic acid cream
- Chronic Sensitivity Test to FS2 cream (Other): Twenty (20) randomized healthy volunteers will be assigned numbers and will have a single testing area identified by permanent marker on either shoulder or upper back. Volunteers will be educated how to apply a pouch of cream to an occlusive, transparent dressing (Tegaderm) and place it on the test site every 24 hours for 30 days. The date and time of first application will be recorded. Baseline urine and serum measurements of drug concentration (presumed absent), as well as complete blood count, liver enzymes, blood urea nitrogen, and creatinine will be taken on Day 0 (the initial enrollment of each part). The volunteers will be seen in follow-up at day 1, day 5, day 15, and day 30.
  Interventions: Drug: Chronic application of kynurenic acid cream

INTERVENTIONS:
Drug: Acute Application of kynurenic acid cream — Pouches containing 0.00% (placebo), 0.15%, 0.25%, 0.4% and 0.5% of FS2 will be randomly applied to an occlusive, transparent dressing (Tegaderm) and applied to each test area. The pouch order will be random, generated by the www.random.org list generator each application. The study team member applying the cream will randomly choose the application sites of different concentrations of the FS2 creams and mark the corresponding cream code name on a separate sheet. This study member will not be evaluating the results and the evaluating study member will be blinded to the randomization. Patients will be evaluated at 24 hours post application for skin reactions and adverse reactions by a blinded observer recorded. Before and after photographs will be taken.
  Other Names: Fibrostop 2 (FS2)
  Arms: Acute Sensitivity Test to FS2 cream
Drug: Chronic application of kynurenic acid cream — Volunteers will be educated how to apply a pouch of cream to an occlusive, transparent dressing (Tegaderm) and place it on the test site every 24 hours for 30 days. The date and time of first application will be recorded. Baseline urine and serum measurements of drug concentration (presumed absent), as well as complete blood count, liver enzymes, blood urea nitrogen, and creatinine will be taken on Day 0 (the initial enrollment of each part). The volunteers will be seen in follow-up at day 1, day 5, day 15, and day 30
  Other Names: Fibrostop 2 (FS2)
  Arms: Chronic Sensitivity Test to FS2 cream

SUMMARY:
Background Scarring typically occurs after trauma, burn injury or surgery. Hypertrophic scarring presents as raised, red and itchy lesions which variably respond to various treatment modalities, such as corticosteroids, pressure garments, laser therapy, the use of silicone sheets and radiotherapy.

Kynurenine, or "Fibrostop 1" (FS1), and its further breakdown products, such as kynurenic acid, or "Fibrostop 2" (FS2), are endogenous products found in many systems and have shown potential in reducing scar formation in animal studies.

The aim of study is to evaluate the safety and tolerability of FS2 cream applied to the skin of healthy human subjects.

DETAILED DESCRIPTION:
Scarring typically occurs after trauma, burn injury or surgery. Hypertrophic scars (scars with excessive amounts of a protein called collagen) and keloids (hypertrophic scars that grow beyond the boundaries of the original wound) are types of abnormal scarring that are termed "dermal fibroproliferative disorders" - disorders of abnormal growth of fibrous tissue in the dermis, a layer in normal skin. These disorders present as raised, red and itchy lesions which variably respond to various treatment modalities, such as corticosteroids, pressure garments, laser therapy, the use of silicone sheets and radiotherapy. Surgical excision of hypertrophic scars or keloids often leads to recurrence resulting in cosmetic deformities and contractures.

In a previous study involving a hypertrophic scar rabbit model, it was found that collagen deposition could be reduced by increasing the activity of a molecule called MMP-1 (matrix metalloproteinase 1), an enzyme inside body cells. The investigators also know from the investigators previous work that a molecule called kynurenine, a breakdown product of amino-acids, can reduce collagen deposition and possibly stimulate MMP production.

Kynurenine is a breakdown product (catabolite) of the essential amino acid tryptophan used in the production of niacin - an organic compound and essential human nutrient found in food. Kynurenine is made by the enzyme indoleamine 2,3-dioxygenase (IDO) which is found in many tissues in response to activation of the immune systen, and also by the enzyme tryptophan dioxygenase, which is found in the liver. Kynurenine is further converted to kynurenic acid, or "Fibrostop 2" (FS2), carry out many functions in the body, including dilating blood vessels during inflammation and regulating the immune response.

The investigators have hypothesized that improved healing outcomes in the investigators rabbit model were due to kynurenine and by-products stimulating MMP, which in turn acted on cells (fibroblasts) to reduce collagen production. This hypothesis lead to a study investigating the effects of topical 0.5% kynurenine cream treatment on MMP-1 and MMP-3 expression in fibrotic rabbit ear wound model. The results showed marked improvement in scar formation suggesting the possible use of kynurenine as an anti-fibrogenic treatment against scarring.

Toxicity, pharmacodynamic, and pharmacokinetic data has been completed, and the investigators institution is now preparing to conduct its first Phase I clinical trial. The investigators objective is to evaluate the safety and tolerability of topically applied FS2 in healthy human subjects by conducting a double-blinded acute and chronic sensitivity study involving patch testing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females between the ages of 18 and 65
* English as a primary language, or English as a second language (ESL) but completely fluent and do not require a translator

Exclusion Criteria:

* Pregnant, or attempting to become pregnant (NB: Pregnancy tests will be administered at the screening and baseline visit.)
* History of chronic skin conditions (e.g: eczema, psoriasis, etc.)
* Use of oral anti-histamines in the past month
* Use of systemic steroids in the past month
* Chronic use of NSAIDs or other anti-inflammatory medications
* Known immunosuppression or immunosuppressive illness
* Known sensitivity to parabens
* Known allergy to the the bandage adhesive
* English as a second language (ESL) and require a translator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Acute skin irritation or local reaction | 24 hours
  After application of various concentrations of the active substance, patients will be evaluated at 24 hours post application for skin reactions and adverse reactions by a blinded observer

SECONDARY OUTCOMES:
Chronic skin irritation or local reaction | 1 month
  After application of various concentrations of the active substance, patients will be evaluated post application for skin reactions and adverse reactions by a blinded observer. The volunteers will be seen in follow-up at day 1, day 5, day 15, and day 30
Chronic exposure serum drug levels | 30 days
  After application of various concentrations of the active substance, patients will have blood taken and analyzed using high performance liquid chromatography. The volunteers will be seen in follow-up at day 1, day 5, day 15, and day 30

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Papp, MD, Principal Investigator — BC Professional Fire Fighters' Burn and Wound Healing Laboratory
Locations (1):
- BCPFF Burn & Wound Healing Lab, Vancouver, British Columbia, Canada